CLINICAL TRIAL: NCT03852446
Title: A Phase 1, Randomized Trial to Evaluate the Pharmacokinetics and Safety of Single Ascending Doses of Indoximod HCl (F2) Tablets (Part 1) and to Compare the Oral Bioavailability of Indoximod Cl (F2) Tablets and Indoximod Free Base Capsule Formulations and the Effect of Food (Part 2) in Healthy Male Volunteers
Brief Title: Single Ascending Dose PK, Oral Bioavailability and Food Effect Study in Healthy Male Volunteers
Acronym: NLG2111
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLG2111
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Indoximod
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose (Experimental)
  Interventions: Drug: Indoximod HCL (F2) tablets; Other: Placebo
- Part 2: Bioavailability and Food Effect (Experimental): 1. Single dose of Indoximod HCL (F2) formulation under fasting conditions
  2. Single dose of Indoximod HCL (F2) formulation under fed conditions
  3. Single dose of Indoximod base formulation under fasting conditions
  Interventions: Drug: Indoximod base formulation; Drug: Indoximod HCL (F2) tablets

INTERVENTIONS:
Drug: Indoximod HCL (F2) tablets — The doses will be ascending per cohort from 600 mg to 2400 mg
  Arms: Part 1: Single Ascending Dose
Drug: Indoximod base formulation — Single oral administration of 1200 mg
  Arms: Part 2: Bioavailability and Food Effect
Other: Placebo — The matching placebo doses will be ascending per cohort from 1 to 4 tablets
  Arms: Part 1: Single Ascending Dose
Drug: Indoximod HCL (F2) tablets — Single oral administration of 1200 mg
  Arms: Part 2: Bioavailability and Food Effect

SUMMARY:
This 2-part study will assess the effect of formulation and food on the pharmacokinetics of Indoximod in healthy volunteers. Part 1 is a randomized single ascending dose study of indoximod salt formulation to characterize the PK profile and determine the safety and tolerability of each dose in healthy male volunteers. Part 2 is an open-label, randomized, 3-period, 3-way crossover study. Participants will receive single doses of Indoximod base or salt formulation, in the fasted or fed state.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months
* BMI within 18 to 30 kg/m2
* Able to speak, read, and understand English or Spanish

Exclusion Criteria:

* Clinically significant cardiac, pulmonary, hepatic or renal disease
* History of substance abuse or alcohol dependence within past 2 years
* Inability to fast for a minimum of 14 hours
* Inability to swallow large capsules/tablets
* Pending legal charges or is on probation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve | up to 20 Days
  Part 2
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | up to 20 Days
  Part 2
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | up to 4 Days
  Part 1

SECONDARY OUTCOMES:
Percentage of patients with adverse events | up to 18 Days
  Part 1
Percentage of patients with adverse events | up to 36 Days
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kennedy, MD, Study Director — NewLink Genetics Inc
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States